CLINICAL TRIAL: NCT06090292
Title: Investigating the Effects of Peripheral Electrical Stimulation in Combination With Low Intensity Focused Ultrasound for Upper Extremity Motor Symptoms in Patients With Parkinson Disease (PD)
Brief Title: Effects of Peripheral Electrical Stimulation With Focused Ultrasound on Motor Symptoms in Parkinson's Patients
Acronym: tbFUS-FES_PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Robert Chen, Senior Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-5740 #3
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will be blind to stimulation condition (sham/active TUS). The assessor for the finger accelerometry will be blind to stimulation condition (sham/active TUS). The UPDRS examination will be video-recorded and blindly assessed by a research team member.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real TUS + Real FES (Experimental): Participants will receive Real TUS using a 2 channel transducer with parameters' of sonication being 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz). The Power of Real tbFUS will be set at 20W. This will be followed by motor point stimulation (MPS) of the right and left hand and forearm muscles i.e. Opponens Pollicis Brevis (OPB), 1st Lumbrical and First Dorsal Interosseous (FDI) muscles triggered in congruence with the voluntary effort of the participant during execution of bilateral functional tasks involving the use of two and three finger pinch grip (e.g.: picking up and moving marbles, ball bearings etc.). Parameters of stimulation will be 40 Hz frequency, 300 microsecs pulse duration, amplitude as per participant tolerance and total stimulation time 30 mins with "ON" time of 4 secs and "OFF" time of 4 secs.
  Interventions: Device: Real TUS; Device: Real FES
- Real TUS +Sham FES (Experimental): Participants will receive Real TUS using a 2 channel transducer with parameters' of sonication being 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz). The Power of Real tbFUS will be set at 20W. This will be followed by motor point stimulation (MPS) of the right and left biceps and long finger flexors triggered in congruence with the voluntary effort of the participant during execution of bilateral functional tasks involving the use of two and three finger pinch grip (e.g.: picking up and moving marbles, ball bearings etc.). Parameters of stimulation will be 40 Hz frequency, 300 microsecs pulse duration, amplitude as per participant tolerance and total stimulation time 30 mins with "ON" time of 4 secs and "OFF" time of 4 secs.
  Interventions: Device: Real TUS; Device: Sham FES
- Sham TUS +Real FES (Experimental): The Sham tbFUS paradigm will consist of 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz), however the ultrasound head will be flipped so that the active side faces away from the head. This will be followed by motor point stimulation (MPS) of the right and left hand and forearm muscles i.e. Opponens Pollicis Brevis (OPB), 1st Lumbrical and First Dorsal Interosseous (FDI) muscles triggered in congruence with the voluntary effort of the participant during execution of bilateral functional tasks involving the use of two and three finger pinch grip (e.g.: picking up and moving marbles, ball bearings etc.). Parameters of stimulation will be 40 Hz frequency, 300 microsecs pulse duration, amplitude as per participant tolerance and total stimulation time 30 mins with "ON" time of 4 secs and "OFF" time of 4 secs.
  Interventions: Device: Real FES; Device: Sham TUS

INTERVENTIONS:
Device: Real TUS — 2 channel transducer from Sonic Concepts will be used to deliver 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz).
  Arms: Real TUS + Real FES; Real TUS +Sham FES
Device: Real FES — Twin Stim Plus EMS stimulator will be used to deliver FES to right and left hand opponens pollicis, first lumbrical and first dorsal interosseous muscles. Parameters of stimulation are 40 Hz frequency, 300 microsecs pulse duration, amplitude as per participant tolerance and total stimulation time 30 mins with "ON" time of 4 secs and "OFF" time of 4 secs.
  Arms: Real TUS + Real FES; Sham TUS +Real FES
Device: Sham TUS — 2 channel transducer from Sonic Concepts will be used to deliver 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz) however the ultrasound head will be flipped so that the active side faces away from the scalp.
  Arms: Sham TUS +Real FES
Device: Sham FES — Twin Stim Plus EMS stimulator will be used to deliver FES to right and left biceps and long finger flexors. Parameters of stimulation are 40 Hz frequency, 300 microsecs pulse duration, amplitude as per participant tolerance and total stimulation time 30 mins with "ON" time of 4 secs and "OFF" time of 4 secs.
  Arms: Real TUS +Sham FES

SUMMARY:
Transcranial Ultrasound Stimulation (TUS) is an emerging non-invasive brain stimulation(NIBS) technique that can be used on both superficial and deep brain targets with a high spatial resolution as small as a few cubic millimeters. Functional Electrical stimulation is a peripheral stimulation technique researched and clinically used to restore motor function following conditions like stroke and Spinal cord injury. To date, there are no studies that have looked at the neuro modulatory effects of combining TUS and FES on motor symptoms in patients with Parkinson's disease. The current study aims to understand the neuromodulatory effects of combining tbFUS to bilateral primary motor cortex (M1) in Parkinsons's disease patients immediately followed by bilateral upper extremity FES of the hand muscles for improving motor symptoms.

DETAILED DESCRIPTION:
There are 3 study visits and for all of them patients will remain in ON dopaminergic medication condition. Each visit will be a minimum of 7 days apart.

Each visit will contain 1 of 3 combinations:

Combination #1: Real TUS +Sham FES; Combination #2: Sham TUS+ Real FES; Combination #3: Real TUS +Real FES

Definition of:

Real TUS: The Real TUS paradigm will consist of 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz). The Power of Real tbFUS will be set at 20W.

Sham TUS: The Sham TUS paradigm will also consist of 120s train of 20ms ultrasound bursts, repeated every 200ms (Pulse Repetition Frequency (PRF)=5Hz), however the ultrasound head will be flipped so that the active side faces away from the head.

Real FES: Motor point stimulation (MPS) of the right and left hand and forearm (Muscles stimulated may include: Opponens Pollicis Brevis (OPB), Flexor Pollicis Brevis, Abductor Pollicis Brevis (APB), 1st Lumbrical, Flexor digitorum superficialis and the First Dorsal Interosseous (FDI)) muscles will be triggered in congruence with the voluntary effort of the Participant during execution of bilateral functional tasks involving the use of two and three finger pinch grip (e.g.: picking up and moving marbles, ball bearings etc.).

Sham FES: Motor point stimulation (MPS) of both right and left Biceps and Finger flexor muscles will be triggered in congruence with the voluntary effort of the participant during execution of bilateral functional tasks involving the use of two and three finger pinch grip (e.g.: picking up and moving marbles, ball bearings etc.).

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years of age
* Confirmed diagnosis of Parkinson's disease
* Stable dopaminergic medication dose for a minimum of 4 weeks (applicable for PD patients only)

Exclusion Criteria:

History of stroke or seizure

* Comorbid dementia
* Scored below 22 on the Montreal Cognitive Assessment (MoCA)
* Has intracranial implant(s) or device(s)
* Has an implanted cardiac pacemaker or implantable cardioverter-defibrillator (ICD)
* Has a previous surgical intervention to treat the movement disorder such as lesioning or a Deep Brain Stimulation system in place.
* Presence of metal implanted in body that is contraindicated in TMS/MRI/peripheral electrical stimulation
* Pregnancy
* Major depression/psychiatric disorder that in the opinion of the Investigator will affect patient's understanding of study procedures and willingness to abide by all procedures during the course of the study
* Is on antipsychotics, anti-depressants, marijuana, or other recreational drugs that affect the nervous system
* Major musculoskeletal or neuromuscular disease or disorder of the hands, wrists and limbs
* Severe Dyskinesia
* Genetic mutations
* Major systemic illness or infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
Averaged 1mV Motor Evoked Potential (MEP) Amplitude recorded from the right and left FDI, APB and ADM | Baseline, immediately after sonication (T0) , T30 (immediately after FES) and T60 (30 minutes after FES).
  To obtain this measurement from both hemispheres, a Transcranial magnetic stimulator's (TMS) power output (expressed as %Maximum Stimulator Output or %MSO) will be adjusted to an intensity that consistently evokes MEP peak-to-peak amplitudes of ~1mV in the right and left FDI when applied to the left primary motor cortex (LM1) and right motor cortex (RM1) respectively, before any neuromodulatory intervention (Pre-I 1mV).

SECONDARY OUTCOMES:
Unified Parkinsons Disease Rating Scale (UPDRS) | Baseline, T30 (immediately after FES) and T60 (30 minutes after FES).
  Change of UPDRS score
Finger tapping task | Baseline, T30 (immediately after FES) and T60 (30 minutes after FES).
  Correlation of the changes in UPDRS scores with the velocity change during finger tapping task as recorded by an accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No